CLINICAL TRIAL: NCT04077645
Title: Examining the Association of Sun Salutations and Aerobic Exercise With Cognition Among Adults With Psychosocial Stress
Brief Title: Yoga and Aerobic Exercise Effects on Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Sean Mullen, PhD, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20067
Record Dates: First submitted 2019-08-22; First posted 2019-09-04 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Stress, Psychological
Keywords: physical activity; walking; moderate intensity; acute intervention
MeSH Terms: conditions — Stress, Psychological; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sun salutations (Experimental): Sun salutations, breathing exercises, and relaxation, at a low to moderate intensity, for 30 minutes.
  Interventions: Behavioral: Sun salutations
- Aerobic exercise (Active Comparator): Walking on a treadmill at low to moderate intensity for 30 minutes.
  Interventions: Behavioral: Aerobic exercise
- Seated rest (attentional control) (Other): Watching educational videos for 30 minutes.
  Interventions: Behavioral: Seated rest

INTERVENTIONS:
Behavioral: Sun salutations — This group will be asked to participate in 25 minutes of low-to-moderate intensity Yoga. This acute session will include engaging in sun salutations, breathing exercises and relaxation. Sun salutations involves performing 10 postures in a particular sequence, and then repeating that sequence. Some of the positions include bending over and touching one's toes, and lying belly-down on the ground and pushing up from ground while arching backwards. The activity will begin as a low intensity activity for the first 5 minutes, and the intensity will be gradually increased. Participants' heart rate will be measured before and after the intervention. The intervention will be delivered by a video displayed on a tablet device. An orientation session in the beginning will familiarize participants with the activity.
  Arms: Sun salutations
Behavioral: Aerobic exercise — This group will be asked to walk on the treadmill for the same amount of time (i.e. 25 minutes) at a moderate intensity (50-70% of their maximum heart rate). Participants will receive an initial 5-minute orientation and then begin at a self-selected speed for the first 5 minutes. Heart rate will be measured and monitored by an undergraduate research assistant. Speed will be increased after 5 minutes if participants have not reached the moderate zone. If participants still have not reached the target heart rate zone by the 10-min mark, the incline of the treadmill will be increased by a 5% grade until the zone is reached.
  Arms: Aerobic exercise
Behavioral: Seated rest — This group will be watching educational videos for the same amount of time as the intervention groups. An orientation session of 5 minutes will be held in the beginning. Participants will be watching videos on general health related topics, such as healthy eating, while being seated in a quiet room, free of distractions.
  Arms: Seated rest (attentional control)

SUMMARY:
The purpose of this acute randomized control study is to assess the feasibility of a low-to-moderate intensity Yoga intervention (i.e. sun salutations), and examine its effect on cognitive functioning, compared to engaging in aerobic activity or seated rest. Participants will include individuals who are currently experiencing symptoms of psychosocial stress or general anxiety.

DETAILED DESCRIPTION:
Eligible participants will be randomized to one of three groups: 1. Sun salutations (Yoga), 2. Aerobic exercise (walking on a treadmill), 3. Seated rest (watching educational videos). Each activity will be 30 minutes in duration. Immediately before and after the 30 minute intervention, participants will undergo psychosocial and cognitive assessments. Prior to the intervention, participant's physical activity will be tracked for one week, via a consumer grade accelerometer.

Baseline and post-intervention testing will include a cognitive battery, psychosocial questionnaires, flexibility testing and physiological measures.

ELIGIBILITY:
Inclusion Criteria:

* Anyone between the ages of 18-45 years
* Anyone with a score of 3 or higher on the Generalized Anxiety Disorder symptom checklist of the Diagnostic and Statistical Manual 5. That is, anyone meeting 3 or more symptoms, on more days of the week than not, for the past 6 months:

  1. Restlessness, feeling keyed up or on edge. 2. Being easily fatigued. 3. Difficulty concentrating or mind going blank. 4. Irritability. 5. Muscle tension. 6. Sleep disturbance (difficulty falling or staying asleep, or restless, unsatisfying sleep).
* Ability to exercise at moderate to vigorous activity levels (defined as 50%-75% of the adjusted age-predicted maximum heart rate)
* Access to a smartphone and willingness to allow research staff to install a mobile activity tracker application (and space to allow for installation)
* Willingness to be randomized into one of three groups

Exclusion Criteria:

* Anyone who is physically active (≥30 minutes, 2 or more times/week, for the last 3 months) and/or a regular practitioner of Yoga or mind-body activities (≥30 minutes, 2 or more times/week, for the last 3 months).
* Anyone with serious chronic medical conditions that would preclude them from participating without a physician present, or anyone with a risk of seizure, or anyone having psychiatric and/or neurological disorders.
* Anyone who does not consent to wearing the Fitbit, or does not have a smartphone that allows us to download an app on their phone.
* Pregnant women.
* Anyone incapable of performing the following movements at a moderate intensity- sitting, standing, kicking, pulling, pushing, bending one's elbows, bending the body forward, bending one's knees, lying down and getting up.
* Anyone with blood pressure of 200/105 or more, and anyone who scores 1 or more on the Physical Activity Readiness Questionnaire
* Anyone refusing or unwilling to be randomized into either of the conditions.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Mullen, PhD, Principal Investigator — University of Illinois at Urbana-Champaign; Madhura Phansikar, MA, Study Director — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Although this is not an NIH-funded study, we will update these records within 1 year of data collection completion per NIH guidelines.
Access Criteria: Data will be accessible on an open site (e.g., Open Science Framework https://osf.io/) with a request to interested parties to engage with the investigative team about any publication of these data in an effort to avoid redundancy. Appropriate authorship crediting investigators involved in the parent study conceptualization, and any consultation regarding data interpretation should be sought by any researchers interested in publishing these data.

REFERENCES:
- See also: Exercise, Technology, and Cognition Laboratory — http://exercisetechlab.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sun Salutations | Aerobic Exercise | Seated Rest (Attentional Control)
Started | 25 | 22 | 24
Completed | 25 | 22 | 24
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sun Salutations | Aerobic Exercise | Seated Rest (Attentional Control) | Total
Number analyzed (Participants) | 25 | 22 | 24 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.19 (8.60) | 28.39 (8.83) | 25.93 (9.16) | 27.84 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 20 | 62
  Male | 3 | 2 | 4 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 11 | 12 | 17 | 40
  African American | 2 | 3 | 3 | 8
  Asian | 10 | 5 | 2 | 17
  Other | 2 | 2 | 2 | 6
N-back Task (Working Memory) [Mean (Standard Deviation); unit: milliseconds] — This is a computerized task measuring the working memory domain of cognition. The task had 3 conditions, namely, 0-back, 1-back and 2-back. Participants are presented with a series of stimuli one after the other. They have to decide whether the stimulus currently presented is the same as the stimulus presented "n" items before. For the 2- back task, they have to decide whether the stimulus matches the stimulus presented 2 earlier. The data presented here is 2-back non-match reaction time, which is the most difficult condition.
  milliseconds | 960.72 (195.07) | 1000 (190.18) | 1002.11 (265.65) | 987.19 (217.88)

OUTCOME MEASURES:

1. Primary Outcome: N-back Task (Working Memory)
Description: This is a computerized task measuring the working memory domain of cognition. The task had 3 conditions, namely, 0-back, 1-back and 2-back. Participants are presented with a series of stimuli one after the other. They have to decide whether the stimulus currently presented is the same as the stimulus presented "n" items before. For the 1-back task, participants have to decide whether the stimulus matches the stimulus presented 1 earlier. For the 2- back task, they have to decide whether the stimulus matches the stimulus presented 2 earlier. Reaction time and accuracy of the response are recorded.
Time Frame: Change from baseline performance on the n-back at 30 minutes
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Sun Salutations | Aerobic Exercise | Seated Rest (Attentional Control)
Number analyzed (Participants) | 25 | 22 | 24
Milliseconds | 827.50 (171.96) | 844.26 (214.36) | 832.60 (217.52)

2. Secondary Outcome: Trail Making Test A and B (Global Cognition)
Description: This is a paper pencil task having 2 parts- Trails A and Trails B, with Trails B being more complex. In Trails A, there are 25 circles on a piece of paper numbered 1-25. Participants have to join these numbers in ascending order, as quickly as they can, without lifting their pencil. In Trails B, the participants have to join 25 circles in an ascending order, but they have to alternate between numbers and letters (1-A-2-B-3-C). Time to complete the task correctly is recorded.
Time Frame: Change from baseline performance at 30 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sun Salutations | Aerobic Exercise | Seated Rest (Attentional Control)
Number analyzed (Participants) | 25 | 22 | 24
seconds | 43.21 (11.12) | 39.18 (8.50) | 40.72 (10.28)

3. Secondary Outcome: Digit Symbol Substitution Test (Processing Speed)
Description: In this task, participants are presented with a code key, in which numbers 1-9 are matched with a unique symbol. Then, they are presented with a sheet of paper having a series of symbols on it. Using the codekey, participants have to read aloud, the numbers that the symbols are associated with, in 2 minutes. The accuracy is recorded.
Time Frame: Change from baseline performance at 30 minutes
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | Sun Salutations | Aerobic Exercise | Seated Rest (Attentional Control)
Number analyzed (Participants) | 25 | 22 | 24
Correct responses | 108.52 (16.73) | 116.23 (12.17) | 120.71 (18.41)

4. Secondary Outcome: State Trait Anxiety Questionnaire
Description: This questionnaire has 20 items for assessing state anxiety. Participants respond on a 4-point scale ("Not at all" to "Very much so"). Composite is calculated by summing the items. Range: 20 (min) - 80 (max). Higher scores indicate greater anxiety.
Time Frame: Change from baseline performance at 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sun Salutations | Aerobic Exercise | Seated Rest (Attentional Control)
Number analyzed (Participants) | 25 | 22 | 24
units on a scale | 30.04 (7.00) | 35.95 (8.93) | 36.00 (9.24)

5. Secondary Outcome: Visual Analog Scale for Stress
Description: Participants have to indicate how stressed they are currently feeling on a scale ranging from 0 (none) to 100 (as bad as it gets). Higher scores mean more stress.
Time Frame: Change from baseline performance at 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sun Salutations | Aerobic Exercise | Seated Rest (Attentional Control)
Number analyzed (Participants) | 25 | 22 | 24
units on a scale | 21.08 (17.22) | 28.82 (25.56) | 38.21 (21.54)

6. Secondary Outcome: Perceived Mental Fatigue
Description: Participants self rate their present moment feelings on a scale from 1 - 5 (1=not true at all, 5=very true) yielding a mean score across all 7 items, with higher scores indicating greater mental fatigue. Range for composite score: 1 (min) - 5 (max).
Time Frame: Change from baseline performance at 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sun Salutations | Aerobic Exercise | Seated Rest (Attentional Control)
Number analyzed (Participants) | 25 | 22 | 24
units on a scale | 1.87 (.59) | 2.01 (.69) | 2.29 (.95)

7. Secondary Outcome: Focus of Attention
Description: Participants are asked to self rate (1 item) their focus of attention while engaged in the previous activity. Responses range from 0 (Internal thoughts) to 10 (external thoughts), with higher scores representing external focus of attention. Range: 0 (min)- 10 (max).
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sun Salutations | Aerobic Exercise | Seated Rest (Attentional Control)
Number analyzed (Participants) | 25 | 22 | 24
units on a scale | 7.84 (1.75) | 2.73 (1.48) | 5.42 (3.02)

8. Secondary Outcome: Feeling Scale
Description: This scale measures how a participant is feeling at the present moment (valence) after a bout of exercise. It is an 11-point one-item measure ranging from +5 (very good) to -5 (very bad). Higher scores represent positive affect. Range: -55 (min) to 55 (max).
Time Frame: Change from baseline performance at 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sun Salutations | Aerobic Exercise | Seated Rest (Attentional Control)
Number analyzed (Participants) | 25 | 22 | 24
units on a scale | 3.68 (1.09) | 2.55 (1.26) | 3.21 (1.64)

9. Secondary Outcome: Heart Rate
Description: Participants' heart rate will be measured using an oxymeter.
Time Frame: Change from baseline performance at 30 minutes
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Sun Salutations | Aerobic Exercise | Seated Rest (Attentional Control)
Number analyzed (Participants) | 25 | 22 | 24
beats per minute | 100.24 (14.40) | 119.27 (6.54) | 69.63 (8.41)

10. Secondary Outcome: Rating of Perceived Exertion
Description: Participants are asked to self rate their feeling of exertion on a 1-item question (11 point scale), ranging from 6 (no exertion) to 20 (maximal exertion), for the activity they were engaged in during the intervention. Range: 6 (min) to 20 (max).
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sun Salutations | Aerobic Exercise | Seated Rest (Attentional Control)
Number analyzed (Participants) | 25 | 22 | 24
units on a scale | 11.24 (2.16) | 11.73 (2.14) | 7.63 (2.39)

11. Secondary Outcome: Rating of Enjoyment and Intervention
Description: Participants will rate their enjoyment in terms of the delivery method and the intervention. This will include questions such as 'Did you like the video instruction for sun salutations?', 'Would you recommend this activity to your family and friends?' Participants had a dichotomous response choice of "yes" or "no". A composite score was calculated as an average across X items. Range of the composite score: 0 to 1. A higher score indicates higher enjoyment.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sun Salutations
Number analyzed (Participants) | 25
units on a scale | .74 (.13)

12. Secondary Outcome: Rating of Technology Ease of Use and Usability
Description: Participants from the yoga group only will rate the technology used to deliver the intervention, in terms of its ease of use and usability. The items are based on the Technology Acceptance Model and will include questions such as 'The Yoga video was clear and understandable.' Response ranges from 1 to 6, and a composite score is reported as an average of the responses. Range of the composite score: 1 (min) - 6 (max). Higher scores represent better technology usability.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sun Salutations
Number analyzed (Participants) | 25
units on a scale | 5.87 (1.03)

ADVERSE EVENTS:
Time Frame: 2 hours
Description: No adverse events occured
Arm/Group | Sun Salutations | Aerobic Exercise | Seated Rest (Attentional Control)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/22 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/22 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT04077645/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT04077645/SAP_001.pdf
  • Informed Consent Form (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT04077645/ICF_002.pdf